CLINICAL TRIAL: NCT01943864
Title: A Phase IIa Study of the MEK Inhibitor GSK1120212 Monotherapy in the Treatment of Gemcitabine Refractory Locally Advanced, Recurrent or Metastatic Biliary Tract Cancers
Brief Title: A Phase IIa Study of the MEK Inhibitor Trametinib Monotherapy in the Treatment of Biliary Tract Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117134
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: pharmacokinetics; second line monotherapy; GSK1120212 (trametinib); MEK inhibitor; locally advanced or metastatic biliary tract cancers
MeSH Terms: conditions — Neoplasms; Biliary Tract Neoplasms | interventions — trametinib; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Trametinib (single tablet) (Experimental): Subjects will receive, trametinib once daily as a single tablet of 2 mg administered orally with eight ounces of water under fasting conditions either one hour before or 2 hours after a meal.
  Interventions: Drug: Trametinib (single tablet)
- Trametinib PK study (multiple tablet) (Experimental): Subjects will receive on Day 1, trametinib as four tablets of 0.5 mg administered orally with eight ounces of water under fasting conditions either one hour before or 2 hours after a meal.
  Interventions: Drug: Trametinib (Multiple tablet)
- Trametinib PK study (single tablet) (Experimental): Subjects will receive Day 2 onwards, trametinib once daily as a single tablet of 2 mg administered orally with eight ounces of water under fasting conditions either one hour before or 2 hours after a meal.
  Interventions: Drug: Trametinib (single tablet)

INTERVENTIONS:
Drug: Trametinib (single tablet) — The drug substance is blended with inert
  Arms: Trametinib (single tablet); Trametinib PK study (single tablet)
Drug: Trametinib (Multiple tablet) — The drug substance is blended with inert
  Arms: Trametinib PK study (multiple tablet)

SUMMARY:
This is a Phase IIa, open-label, single-arm, multi-center study to evaluate the efficacy and safety of orally administered MEK inhibitor trametinib as the second line in subjects with advanced or metastatic biliary tract cancers (BTC) in Japanese population. The primary endpoint of this study is 12 week non-progressive disease (PD) rate defined as the percentage of subjects without progression at Week 12. As a sub-study, pharmacokinetics (PK) of four tablets of 0.5 milligram (mg) tablet, or one tablet of 2 mg tablet to achieve 2 mg daily regimen will be assessed to evaluate the pharmacokinetics of trametinib in Japanese population.

Eligible subjects will be randomized to receive trametinib at the recommended Phase II dose of 2 mg every day as one 2 mg tablet or four 0.5 mg tablets on Day 1. From Day 2 until disease progression or withdrawal from the study treatment, all subjects will receive one tablet of 2 mg trametinib . Disease assessment will be performed every 8 week. Translational research is also planned to evaluate the potential blood or tumor tissue-derived biomarkers for biological activity, and sensitivity or resistance to treatment with trametinib .

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age 20 years or older inclusive, at the time of signing the informed consent.
* Japanese patients with histologically or cytologically confirmed cholangiocarcinoma (intra- or extrahepatic) or gallbladder cancer or ampulla of Vater cancer are eligible for which all of the following criteria have to be met: Nonresectable, recurrent, and/or metastatic disease.
* Disease progression after up to two lines of systemic chemotherapies including no more than one line of gemcitabine-based chemotherapy. Note: Systemic therapy in adjuvant setting is not allowed as prior therapy.
* More than 21 days have elapsed since any prior anti-tumor therapy.
* At least one of the tumor samples for archived tissue at initial diagnosis or archived tissue at recent progression or fresh biopsy at recent progression (collect within 21 days from randomization if none of the archived tissues are available) is available prior to randomization to provide for translational research.
* Measurable disease, i.e. presenting with at least one measurable lesion per the RESIST 1.1.
* Performance status score of ≤1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Estimated life expectancy of at least 12 weeks.
* All prior treatment- related toxicities must be common terminology criteria for adverse events (CTCAE) (Version 4.0) ≤ Grade 1 (except alopecia) at the time of randomization.
* Negative for hepatitis C virus (HCV) test, hepatitis B surface (HBs) antigen, hepatitis virus Bc (HBc) antibody, and HBs antibody. HBs antigen-negative subjects who test positive for both HBc antibody and HBs antibody or either of them may be eligible when their HBV DNA quantification result is negative.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study treatment and agree to use effective contraception throughout the treatment period, and for 4 months after the last dose of study treatment.
* Adequate baseline organ function for haematological, hepatic, renal, cardiac systems.

Exclusion Criteria:

* History of another malignancy.
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Radiotherapy completed within 2 weeks prior to randomization.
* History of interstitial lung disease or pneumonitis.
* Having a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 28 days prior to randomization and/or chemotherapy without the potential for delayed toxicity within 21days prior to randomization.
* Any prior use of any MEK inhibitors (including but not limited to trametinib, AZD6244 (selumetinib), RDEA119).
* Current use of a prohibited medication.
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression.
* Known Human Immunodeficiency Virus (HIV) infection. History or evidence of cardiovascular risk including a QT interval corrected for heart rate using the Bazett's formula (QTcB) interval >480 msec, history or evidence of current clinically significant uncontrolled arrhythmias, history of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization, history or evidence of current > or = Class II congestive heart failure as defined by New York Heart Association, treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy, subjects with intra-cardiac defibrillators or permanent pacemakers.
* Known cardiac metastases.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09-19; Primary Completion 2014-07-01 (Actual); Study Completion 2016-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Ikeda M, Ioka T, Fukutomi A, Morizane C, Kasuga A, Takahashi H, Todaka A, Okusaka T, Creasy CL, Gorman S, Felitsky DJ, Kobayashi M, Zhang F, Furuse J. Efficacy and safety of trametinib in Japanese patients with advanced biliary tract cancers refractory to gemcitabine. Cancer Sci. 2018 Jan;109(1):215-224. doi: 10.1111/cas.13438. Epub 2017 Dec 9. PMID 29121415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced or metastatic biliary tract cancers (BTC) with unresectable measurable disease which had progressed after one gemcitabine-based chemotherapy were included in the study.
Pre-assignment Details: Participants meeting eligibility criteria received GSK1120212 treatment.
Groups:
- GSK1120212 2 mg: Participants received GSK1120212 at 2 milligram (mg), either as four tablets of 0.5 mg or one tablet of 2 mg at Day 1. At Day 2 and for the remaining study period, participants received continuous daily dosing of one tablet of 2 mg GSK1120212 once-daily until disease progression or death or until study treatment stopping criteria was met.
Period: Overall Study
Arm/Group | GSK1120212 2 mg
Started | 20
Completed | 20 (Death or 1 year from randomization after progression was considered completion; 20 participants died)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Indicated Non-progressive Disease as Assessed by Investigator Per Response Evaluation Criteria In Solid Tumor Version 1.1 (RECIST 1.1) at Week 12
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions; Stable Disease(SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Progressive Disease(PD), At least a 20% increase in the sum of the diameters of target lesions. Non-PD = CR + PR + SD.
Time Frame: Up to Week 12
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 2
  Non-CR/Non-PD | 0
  Progressive Disease (PD) | 3
  Not Evaluable (NE) | 0
  Progressive Disease before week 12 | 12
  Censored before week 12 | 3
  CR+PR+SD+Non-CR/Non-PD | 2
Statistical Analysis 1: Comparison: GSK1120212 2 mg; Test type: Superiority or Other; p = 0.976, Exact Binomial Test; non PD rate at Week 12 = 10, 95% CI 2-sided [1.2 to 31.7]

2. Primary Outcome: Number of Participants With Indicated Non-progressive Disease as Assessed by Independent Radiologist Per Response Evaluation Criteria In Solid Tumor Version 1.1 (RECIST 1.1) at Week 12
Description: Twelve week non-progressive disease (PD) at Week 12 was evaluated by computed tomography. Non- PD was calculated as the sum of complete response (CR), partial response (PR), and stable disease (SD).
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 3
  Non-CR/Non-PD | 0
  Progressive Disease (PD) | 2
  Not Evaluable (NE) | 0
  Progressive Disease before week 12 | 11
  Censored before week 12 | 4
  CR+PR+SD+Non-CR/Non-PD | 3
Statistical Analysis 1: Comparison: GSK1120212 2 mg; Test type: Superiority or Other; p = 0.909, Exact Binomial Test; non PD rate at Week 12 = 15, 95% CI 2-sided [3.2 to 37.9]

3. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect or Protocol-Specific SAEs
Time Frame: until 26-Feb-2016
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Any AE | 20
  Any SAE | 13

4. Secondary Outcome: Expression of Interstitial Lung Disease Marker KL-6
Description: Interstitial lung disease markers KL-6 assessments were carried out at Baseline (Day 1), Week 12, Week 20, Week 24, Week 28, Week 32, and Week 36
Time Frame: From Baseline up to Week 36
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period. Only those participants with analyzable data at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: Units/milliliter (U/mL)
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Units/milliliter (U/mL)
  Baseline, n=20 | 484.36 (568.071)
  Week 12, n=3 | 2664.00 (3786.380)
  Week 20, n=1 | 152.00 (NA) — SD is not applicable, as there was only one participant analyzable
  Week 24, n=1 | 207.00 (NA) — SD is not applicable, as there was only one participant analyzable
  Week 28, n=2 | 313.00 (162.635)
  Week 32, n=1 | 226.00 (NA) — SD is not applicable, as there was only one participant analyzable
  Week 36, n=1 | 237.00 (NA) — SD is not applicable, as there was only one participant analyzable

5. Secondary Outcome: Expression of Interstitial Lung Disease Marker Surfactant Protein D
Description: Interstitial lung disease marker Surfactant Protein D assessments were carried out at Baseline (Day 1), Week 12, and Week 28
Time Frame: Baseline, Week 12, and Week 28
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period. Only those participants with analyzable data at the indicated time point were assessed (represented by n=x).
Measure: Mean (Standard Deviation); unit: Micrograms per litre (µ/L)
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Micrograms per litre (µ/L)
  Baseline, n=17 | 155.98 (428.071)
  Week 12, n=2 | 512.00 (507.703)
  Week 28, n=1 | 77.40 (NA) — SD is not applicable, as there was only one participant analyzable.

6. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Clinical Chemistry Grade Shifts From Baseline
Description: Shift from baseline was calculated as the post baseline value minus the baseline value for albumin, alkalaine phosphatase (AP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, creatine kinase (CK), creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, and phosphate. A Worst Post Baseline (WPB) grade shift is defined as the worst change that occurred at any measured timepoint during the treatment period. Grading was determined by the NCI Common Terminology Criteria for Adverse Events Version 3.0 (NCI-CTCAE). Participants with missing baseline grade were designated a baseline grade of 0.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Albumin, WPB, Any grade increase, n=20 | 13
  Albumin, WPB, Increase to grade 3, n=20 | 1
  Albumin, WPB, Increase to grade 4, n=20 | 0
  AP, WPB, Any grade increase, n=20 | 9
  AP, WPB, Increase to grade 3, n=20 | 2
  AP, WPB, Increase to grade 4, n=20 | 0
  ALT, WPB, Any grade increase, n=20 | 9
  ALT, WPB, Increase to grade 3, n=20 | 3
  ALT, WPB, Increase to grade 4, n=20 | 0
  AST, WPB, Any grade increase, n=20 | 13
  AST, WPB, Increase to grade 3, n=20 | 2
  AST, WPB, Increase to grade 4, n=20 | 0
  Bilirubin, WPB, Any grade increase, n=20 | 4
  Bilirubin, WPB, Increase to grade 3, n=20 | 2
  Bilirubin, WPB, Increase to grade 4, n=20 | 1
  CK, WPB, Any grade increase, n=2 | 1
  CK, WPB, Increase to grade 3, n=2 | 0
  CK, WPB, Increase to grade 4, n=2 | 0
  Creatinine, WPB, Any grade increase, n=20 | 4
  Creatinine, WPB, Increase to grade 3, n=20 | 0
  Creatinine, WPB, Increase to grade 4, n=20 | 0
  Hypercalcemia, WPB, Any grade increase, n=20 | 1
  Hypercalcemia, WPB, Increase to grade 3, n=20 | 0
  Hypercalcemia, WPB, Increase to grade 4, n=20 | 0
  Hyperglycemia, WPB, Any grade increase, n=20 | 10
  Hyperglycemia, WPB, Increase to grade 3, n=20 | 1
  Hyperglycemia, WPB, Increase to grade 4, n=20 | 0
  Hyperkalemia, WPB, Any grade increase, n=20 | 1
  Hyperkalemia, WPB, Increase to grade 3, n=20 | 0
  Hyperkalemia, WPB, Increase to grade 4, n=20 | 0
  Hypermagnesemia, WPB, Any grade increase, n=20 | 1
  Hypermagnesemia, WPB, Increase to grade 3, n=20 | 0
  Hypermagnesemia, WPB, Increase to grade 4, n=20 | 0
  Hypernatremia, WPB, Any grade increase, n=20 | 0
  Hypernatremia, WPB, Increase to grade 3, n=20 | 0
  Hypernatremia, WPB, Increase to grade 4, n=20 | 0
  Hypocalcemia, WPB, Any grade increase, n=20 | 0
  Hypocalcemia, WPB, Increase to grade 3, n=20 | 0
  Hypocalcemia, WPB, Increase to grade 4, n=20 | 0
  Hypoglycemia, WPB, Any grade increase, n=20 | 1
  Hypoglycemia, WPB, Increase to grade 3, n=20 | 0
  Hypoglycemia, WPB, Increase to grade 4, n=20 | 0
  Hypokalemia, WPB, Any grade increase, n=20 | 1
  Hypokalemia, WPB, Increase to grade 3, n=20 | 1
  Hypokalemia, WPB, Increase to grade 4, n=20 | 0
  Hypomagnesemia, WPB, Any grade increase, n=20 | 0
  Hypomagnesemia, WPB, Increase to grade 3, n=20 | 0
  Hypomagnesemia, WPB, Increase to grade 4, n=20 | 0
  Hyponatremia, WPB, Any grade increase, n=20 | 1
  Hyponatremia, WPB, Increase to grade 3, n=20 | 0
  Hyponatremia, WPB, Increase to grade 4, n=20 | 0
  Phosphate, WPB, Any grade increase, n=20 | 2
  Phosphate, WPB, Increase to grade 3, n=20 | 0
  Phosphate, WPB, Increase to grade 4, n=20 | 0

7. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Coagulation Grade Shifts From Baseline
Description: Shift from baseline was calculated as the post baseline value minus the baseline value for activated partial thromboplastin time (APTT) and prothrombin time (PT). A Worst Post Baseline (WPB) grade shift is defined as the worst change that occurred at any measured timepoint during the treatment period. Grading was determined by the NCI Common Terminology Criteria for Adverse Events Version 3.0 (NCI-CTCAE). Participants with missing baseline grade were designated a baseline grade of 0.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  APTT, WPB, Any grade increase, n=18 | 1
  APTT, WPB, Increase to grade 3, n=18 | 0
  APTT, WPB, Increase to grade 4, n=18 | 0
  PT, WPB, Any grade increase, n=18 | 5
  PT, WPB, Increase to grade 3, n=18 | 0
  PT, WPB, Increase to grade 4, n=18 | 0

8. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Hematology Grade Shifts From Baseline
Description: Shift from baseline was calculated as the post baseline value minus the baseline value for hemoglobin, lymphocytes, neutrophils, platelets, and leukocytes. A Worst Post Baseline (WPB) grade shift is defined as the worst change that occurred at any measured timepoint during the treatment period. Grading was determined by the NCI Common Terminology Criteria for Adverse Events Version 3.0 (NCI-CTCAE). Participants with missing baseline grade were designated a baseline grade of 0.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Hemoglobin, WPB, Any grade increase, n=20 | 7
  Hemoglobin, WPB, Increase to grade 3, n=20 | 3
  Hemoglobin, WPB, Increase to grade 4, n=20 | 0
  Lymphocytes, WPB, Any grade increase, n=20 | 6
  Lymphocytes, WPB, Increase to grade 3, n=20 | 1
  Lymphocytes, WPB, Increase to grade 4, n=20 | 0
  Neutrophils, WPB, Any grade increase, n=20 | 3
  Neutrophils, WPB, Increase to grade 3, n=20 | 0
  Neutrophils, WPB, Increase to grade 4, n=20 | 0
  Platelets, WPB, Any grade increase, n=20 | 2
  Platelets, WPB, Increase to grade 3, n=20 | 0
  Platelets, WPB, Increase to grade 4, n=20 | 1
  Leukocytes, WPB, Any grade increase, n=20 | 2
  Leukocytes, WPB, Increase to grade 3, n=20 | 0
  Leukocytes, WPB, Increase to grade 4, n=20 | 0

9. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Clinical Chemistry Measurements With Respect to the Normal Range
Description: Change from baseline was calculated as the post baseline value minus the baseline value for cancer antigen 19-9 (CA 19-9), chloride, lactate dehydrogenase (LDH), and urea. A Worst Post Baseline (WPB) change is defined as the worst change that occurred at any measured timepoint during the treatment period. Measurements were designated as either Decreased to Low (DTL) or Increased to High (ITH) or Change to Normal/No Change (CN/NC). Participants with missing baseline measurements or visit measurements were considered to be missing. Participants were counted twice if the participant Decreased to Low and Increased to High.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  CA 19-9,WPB,DTL,n=20 | 0
  CA 19-9,WPB,CN/NC,n=20 | 18
  CA 19-9,WPB,ITH,n=20 | 2
  Chloride,WPB,DTL,n=20 | 2
  Chloride,WPB,CN/NC,n=20 | 16
  Chloride,WPB,ITH,n=20 | 2
  LDH,WPB,DTL,n=20 | 1
  LDH,WPB,CN/NC,n=20 | 5
  LDH,WPB,ITH,n=20 | 14
  Urea,WPB,DTL,n=20 | 2
  Urea,WPB,CN/NC,n=20 | 15
  Urea,WPB,ITH,n=20 | 3

10. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Prothrombin Time Measurements With Respect to the Normal Range
Description: Change from baseline was calculated as the post baseline value minus the baseline value for prothrombin time (PT). A Worst Post Baseline (WPB) change is defined as the worst change that occurred at any measured timepoint during the treatment period. Measurements were designated as either Decreased to Low (DTL) or Increased to High (ITH) or Change to Normal/No Change (CN/NC). Participants with missing baseline measurements or visit measurements were considered to be missing. Participants were counted twice if the participant Decreased to Low and Increased to High.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 10
Participants
  PT,WPB,DTL,n=11 | 0
  PT,WPB,CN/NC,n=11 | 8
  PT,WPB,ITH,n=11 | 3

11. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Hematology Measurements With Respect to the Normal Range
Description: Change from baseline was calculated as the post baseline value minus the baseline value for basophils, eosinophils, and monocytes. A Worst Post Baseline (WPB) change is defined as the worst change that occurred at any measured timepoint during the treatment period. Measurements were designated as either Decreased to Low (DTL) or Increased to High (ITH) or Change to Normal/No Change (CN/NC). Participants with missing baseline measurements or visit measurements were considered to be missing. Participants were counted twice if the participant Decreased to Low and Increased to High.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Basophils,WPB,DTL,n=20 | 0
  Basophils,WPB,CN/NC,n=20 | 19
  Basophils,WPB,ITH,n=20 | 1
  Eosinophils,WPB,DTL,n=20 | 4
  Eosinophils,WPB,CN/NC,n=20 | 12
  Eosinophils,WPB,ITH,n=20 | 5
  Monocytes,WPB,DTL,n=20 | 2
  Monocytes,WPB,CN/NC,n=20 | 14
  Monocytes,WPB,ITH,n=20 | 5

12. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Carcinoembryonic Antigen Measurements With Respect to the Normal Range
Description: Change from baseline was calculated as the post baseline value minus the baseline value for carcinoembryonic antigen (CEA). A Worst Post Baseline (WPB) change is defined as the worst change that occurred at any measured timepoint during the treatment period. Measurements were designated as either Decreased to Low (DTL) or Increased to High (ITH) or Change to Normal/No Change (CN/NC). Participants with missing baseline measurements or visit measurements were considered to be missing. Participants were counted twice if the participant Decreased to Low and Increased to High.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  CEA,WPB,DTL,n=19 | 0
  CEA,WPB,CN/NC,n=19 | 17
  CEA,WPB,ITH,n=19 | 2

13. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Body Temperature
Description: Body temperature was categorized as Decrease to <=35; Change to Normal or No Change and Increase to >=38. Change from baseline was calculated as the post baseline value minus the baseline value. A Worst Post Baseline (WPB) change is defined as the worst change that occurred at any measured timepoint during the treatment period. Participants with missing baseline measurements or visit measurements were considered to be missing.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  WPB, Decrease to <=35, n=20 | 0
  WPB, Change to normal or no change , n=20 | 18
  WPB, Increase to >=38, n=20 | 2

14. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Blood Pressure
Description: Systolic and diastolic blood pressure was measured after sitting for at least 5 minutes. Systolic blood pressure (SBP) was categorized as: Grade 0 (<120), Grade 1 (>=120-<140), Grade 2 (>=140-<160) and Grade 3 (>=160). Diastolic blood pressure (DBP) was categorized as Grade 0 (<80), Grade 1 (>=80-<90), Grade 2 (>=90-<100), and Grade 3 (>=100). Change from baseline was calculated as the post baseline value minus the baseline value. A Worst Post Baseline (WPB) change is defined as the worst change that occurred at any measured timepoint during the treatment period. Participants with missing baseline measurements or visit measurements were considered to be missing.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  SBP, WPB, Any grade increase, n=20 | 8
  SBP, WPB, Increase to grade 2, n=20 | 4
  SBP, WPB, Increase to grade 3, n=20 | 0
  DBP, WPB, Any grade increase, n=20 | 8
  DBP, WPB, Increase to grade 2, n=20 | 3
  DBP, WPB, Increase to grade 3, n=20 | 2

15. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Pulse Rate
Description: Pulse rate was categorized as Decrease to <60, Change to Normal or No Change, and Increase to >100. Change from baseline was calculated as the post baseline value minus the baseline value. A Worst Post Baseline (WPB) change is defined as the worst change that occurred at any measured timepoint during the treatment period. Participants with missing baseline measurements or visit measurements were considered to be missing.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  PR, WPB, Decrease to <60, n=20 | 0
  PR, WPB, Change to normal or no change, n=20 | 19
  PR, WPB, Increase to >100, n=20 | 1

16. Secondary Outcome: Change From Baseline in Oxygen Saturation (SpO2)
Description: Oxygen Saturation was measured at Baseline (Day 1), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32 and Week 36. For records occurring after baseline, change from baseline was calculated as the post baseline value minus the baseline value. When either the baseline or visit value was missing, the change from baseline was considered to be missing.
Time Frame: From Baseline up to Week 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent oxygen saturation
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Percent oxygen saturation
  Week 4, n=20 | 0.5 (1.15)
  Week 8, n=11 | 0.1 (2.34)
  Week 12, n=5 | 0.4 (1.82)
  Week 16, n=2 | 1.0 (1.41)
  Week 20, n=2 | 0.0 (1.41)
  Week 24, n=2 | 0.5 (2.12)
  Week 28, n=2 | -2.0 (4.24)
  Week 32, n=1 | 2.0 (NA) — SD is not applicable, as there was only one participant analyzable
  Week 36, n=1 | 2.0 (NA) — SD is not applicable, as there was only one participant analyzable

17. Secondary Outcome: Number of Participants With Progression-Free Survival as Assessed by Investigator
Description: Progression-Free Survival (PFS) is defined as the interval of time (in weeks) between the date of randomization and the earlier of the date of disease progression and the date of death due to any cause. Disease progression was based on the assessments by the Investigator. If a participant received subsequent anti-cancer therapy prior to the date of documented progression or death, PFS in the participant was censored at the last adequate assessment prior the initiation of the new anti-cancer therapy. Otherwise, if a participant did not have a documented date of progression or death, PFS in the participant was censored at the last adequate assessment.
Time Frame: Up to Week 37
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Progression or Death | 18
  Censored, follow-up ended | 2
  Censored, follow-up ongoing | 0
Statistical Analysis 1: Comparison: GSK1120212 2 mg; Test type: Superiority or Other; Median PFS = 10.6, 95% CI 2-sided [4.6 to 12.1] — Lower and upper limits and estimation value are in terms of weeks

18. Secondary Outcome: Number of Participants With Progression-Free Survival as Assessed by Independent Radiologist
Description: Progression-Free Survival (PFS) is defined as the interval of time (in weeks) between the date of randomization and the earlier of the date of disease progression and the date of death due to any cause. Disease progression was based on the assessments by the independent radiologist. If a participant received subsequent anti-cancer therapy prior to the date of documented progression or death, PFS in the participant was censored at the last adequate assessment prior the initiation of the new anti-cancer therapy. Otherwise, if a participant did not have a documented date of progression or death, PFS in the participant was censored at the last adequate assessment.
Time Frame: Up to Week 37
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Progression or Death | 16
  Censored, follow-up ended | 4
  Censored, follow-up ongoing | 0
Statistical Analysis 1: Comparison: GSK1120212 2 mg; Test type: Superiority or Other; Median PFS = 10.6, 95% CI 2-sided [4.6 to 12.7] — Lower and upper limits and estimation value are in terms of weeks

19. Secondary Outcome: Number of Participants With Overall Survival
Description: Overall Survival (OS) is defined as the interval of time (in weeks) between the date of randomization and the date of death due to any cause. For participants that did not die, time of death was censored at the date of last contact. The date of death was taken from that recorded on the Record of Death page. Death on study due to any cause was included. One year OS was calculated from Kaplan-Meier estimates.
Time Frame: Up to Week 39
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Death (event) at or prior to 1 year | 16
  Censored, Alive with less than 1 year follow-up | 0
  Censored, Alive with more than 1 year follow-up | 4
  Censored, Died after 1 year | 0
Statistical Analysis 1: Comparison: GSK1120212 2 mg; Test type: Superiority or Other; Overall Survival = 20, 95% CI 2-sided [6.2 to 39.3]

20. Secondary Outcome: Number of Participants With Overall Response Rate as Assessed by Investigator Per RECIST 1.1 Criteria
Description: Overall Response Rate (ORR) is defined as the number of participants achieving a confirmed CR or PR per RECIST 1.1 criteria from the start of treatment until disease progression or the start of new anti-cancer therapy. ORR was based on responses from the Investigator assessment of best overall response, the best overall response is the best response recorded from the start of the treatment until disease progression/recurrence. ORR is calculated as CR + PR.
Time Frame: Up to Week 37
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Complete response (CR) | 0
  Partial response (PR) | 0
  CR + PR | 0
Statistical Analysis 1: Comparison: GSK1120212 2 mg; Test type: Superiority or Other; ORR = 0, 95% CI 2-sided [0 to 16.8]

21. Secondary Outcome: Number of Participants With Overall Response Rate as Assessed by Independent Radiologist Per RECIST 1.1 Criteria
Description: Overall Response Rate (ORR) is defined as the number of participants achieving a confirmed CR or PR per RECIST 1.1 criteria from the start of treatment until disease progression or the start of new anti-cancer therapy. ORR was based on responses from the Independent Radiologist assessment of best overall response, the best overall response is the best response recorded from the start of the treatment until disease progression/recurrence. ORR is calculated as CR + PR.
Time Frame: Up to Week 37
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 20
Participants
  Complete response (CR) | 0
  Partial response (PR) | 1
  CR + PR | 1
Statistical Analysis 1: Comparison: GSK1120212 2 mg; Test type: Superiority or Other; ORR = 5, 95% CI 2-sided [0.1 to 24.9]

22. Secondary Outcome: Number of Participants With Investigator-Assessed Time to Response
Description: Time to response (TTR) event was defined as achievement of a confirmed CR or PR, as the time from date of randomization until date of first documented evidence of CR or PR (whichever status is recorded first). If a participant received subsequent anti-cancer therapy prior to the date of documented progression or death, progression free survival (PFS) in the participant was censored at the last adequate assessment prior the initiation of the new anti-cancer therapy. Otherwise, if a participant did not have a documented date of progression or death, PFS in the participant was censored at the last adequate assessment.
Time Frame: Up to Week 37
Population: ITT Population.
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 0

23. Secondary Outcome: Number of Weeks Until Time to Response Assessed With Independent Radiologist
Description: Time to response (TTR) event was defined as achievement of a confirmed CR or PR, as the time from date of randomization until date of first documented evidence of CR or PR (whichever status is recorded first). If a participant received subsequent anti-cancer therapy prior to the date of documented progression or death, progression free survival (PFS) in the participant was censored at the last adequate assessment prior the initiation of the new anti-cancer therapy. Otherwise, if a participant did not have a documented date of progression or death, PFS in the participant was censored at the last adequate assessment. Only 1 participant reached PR therefore estimated time to response cannot be presented. The time to response for this patient is presented as the actual number of weeks to PR.
Time Frame: Up to Week 37
Population: ITT Population. Only 1 participant reached PR therefore estimated time to response cannot be presented. The time to response for this patient is presented as the actual number of weeks to PR.
Measure: Number; unit: Weeks
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 1
Weeks | 20.1

24. Secondary Outcome: Number of Participants With Investigator-Assessed Duration of Response
Description: Duration of response was summarized for participants with a confirmed CR or PR and is defined as the time (in weeks) from the initial response (CR/PR) to first documented disease progression or death due to any cause. If a participant received subsequent anti-cancer therapy prior to the date of documented progression or death, PFS in the participant was censored at the last adequate assessment prior the initiation of the new anti-cancer therapy. Otherwise, if a participant did not have a documented date of progression or death, PFS in the participant was censored at the last adequate assessment.
Time Frame: Up to Week 37
Population: ITT Population with a time to response event.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 1
Participants
  Progression or Death (event) | 0
  Censored, follow-up ended | 1
  Censored, follow-up ongoing | 0

25. Secondary Outcome: Number of Participants With Independent Radiologist Assessed Duration of Response
Description: as for outcome 24
Time Frame: Up to Week 37
Population: ITT Population with a time to response event. Only 1 participant reached PR therefore estimated time to response cannot be presented. At the data cut off, this patient is censored. Therefore, the observed value of duration of response is unknown.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg
Number analyzed (Participants) | 1
Participants
  Progression or Death (event) | 0
  Censored, follow-up ended | 1
  Censored, follow-up ongoing | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the time the first dose of study treatment until 30 days following discontinuation of study treatment.
Description: SAEs and non-serious AEs are reported for members of the Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | GSK1120212 2 mg
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 2 mg (N=20)
Cholangitis (Hepatobiliary disorders) | 4
Bile duct stenosis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Biliary tract infection (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Chorioretinopathy (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Blood bilirubin increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Presyncope (Nervous system disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Amylase increased (Investigations) | 1
Weight decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 2 mg (N=20)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15
Rash (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 3
Anal haemorrhage (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 6
Malaise (General disorders) | 5
Oedema (General disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Pharyngitis (Infections and infestations) | 4
Paronychia (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Blood creatine phosphokinase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 3
C-reactive protein increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Vision blurred (Eye disorders) | 2
Growth of eyelashes (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangitis (Hepatobiliary disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 1
Insomnia (Psychiatric disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 3
Ear pain (Ear and labyrinth disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Duodenal obstruction (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Glocose tolerance impaired (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Angular cheilitis (Infections and infestations) | 1
Cataract (Eye disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.